CLINICAL TRIAL: NCT04948047
Title: Assessment of the Efficacy of Breath Test Combined With Computed Tomography for Diagnoses of Pulmonary Nodules.
Brief Title: Breath Combined With CT for Diagnoses of Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Jiangsu Cancer Institute & Hospital (Other); Beijing Breatha Biological Technology Co., Ltd, Beijing (Unknown)
Responsible Party: Principal Investigator, Mantang Qiu, MD, PhD, Research Assistant, Peking University People's Hospital
Other Study IDs: 2021PHB150-001
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer; Pulmonary Nodule, Multiple
Keywords: volatile organic compound; pulmonary nodules; predictive model; computed tomography; HPPI-TOFMS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Multiple Pulmonary Nodules | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Volatile organic compound (VOC) in exhalation collected with air bags.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant pulmonary nodules: Patients with pulmonary nodule diagnosed as malignant cancer by pathological examinations after surgical resection.
  Interventions: Diagnostic Test: Pathological examinations as the golden diagnosis criteria; Diagnostic Test: Breath test combined with computed tomography
- Benign pulmonary nodules: Patients with pulmonary nodule diagnosed as benign disease by pathological examinations after surgical resection.
  Interventions: Diagnostic Test: Pathological examinations as the golden diagnosis criteria; Diagnostic Test: Breath test combined with computed tomography

INTERVENTIONS:
Diagnostic Test: Pathological examinations as the golden diagnosis criteria — Pathological diagnosis, as the golden standard for diagnosing pulmonary nodules, is achieved by two experienced pathologists and validated by the third senior pathologist.
Diagnostic Test: Breath test combined with computed tomography — Exhaled breath of each participant will be collected with Tedlar bags. The volatile organic compounds will be detected by a high-resolution high-pressure photon ionization time-of-ﬂight mass spectrometry (HPPI-TOFMS).
  The Imaging markers of pulmonary nodules, including the size, three-dimensional shape, and appearance characteristics, are derived from the chest computed tomography within 2 weeks before surgery resection.

SUMMARY:
Pulmonary nodules diagnosis using breath test of volatile organic compound (VOC) is in its infancy. The accuracy of VOC analysis in diagnosing malignant pulmonary nodules varies cross the published studies. The diagnosis accuracy of VOC alone is generally poor. We speculate that the accuracy of diagnosing malignant pulmonary nodules will be improved by combining breath test with chest computed tomography (CT). This study aims to establish a predictive model of malignant pulmonary nodule using bio-markers from exhaled breath and image-markers from chest CT with retrospective data from multi centers. The sensitivity, specificity and accuracy of the model will be validated prospectively.

DETAILED DESCRIPTION:
Endogenous volatile organic compounds (VOCs) can be derived from many different metabolic pathways. VOCs can be transported to the alveoli through the blood circulation and expelled by exhalation. Changes in VOCs production, clearance, and alterations in lung air-blood exchange functions can lead to aberrant VOCs profiles in the exhaled breath. Testing exhaled breath has the advantages of being completely non-invasive and easy to collect, and has been considered as a perfect approach for disease diagnoses and therapeutic monitoring. Many clinical studies have found that VOCs in exhaled breath are closely related to disease status. Specific VOCs alterations have been identified in many tumors, especially lung cancer. Pulmonary nodules diagnosis using breath test of volatile organic compound (VOC) is in its infancy. The accuracy of VOC analysis in diagnosing malignant pulmonary nodules varies cross the published studies. The diagnosis accuracy of VOC alone is generally poor. We speculate that the accuracy of diagnosing malignant pulmonary nodules will be improved by combining VOC analysis with chest computed tomography.

In this study, we use a highly sensitive mass spectrometry to detect exhaled VOCs of patients with pulmonary nodules. The chest CT will be used for detecting the imaging characteristics of pulmonary nodules. The pathological diagnosis of pulmonary nodules after surgical resections is selected as golden standard.

This study aims to establish a predictive model of malignant pulmonary nodule using bio-markers from breath test and image-markers from chest CT with retrospective data from multi centers. The sensitivity, specificity and accuracy of the model will be varied prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old;
2. Pulmonary nodules with planned surgical resection;
3. Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

1. Preoperative radiotherapy, chemotherapy, targeted therapy or other anti-tumor therapy
2. The lack of chest computed tomography within two weeks before surgery
3. A history of malignant disease within 5 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To establish pulmonary nodule diagnosis model of breath test combined with computed tomography, we reviewed the prospective database established during the study of NCT04419207 for participant recruitment. 200 participants with malignant pulmonary nodules and 200 patients with benign pulmonary nodules will be included for establishing the diagnosis model.
  To validate the efficacy of the established model in distinguishing malignant pulmonary nodules from benign nodules, we will prospectively recruit 500 patients with pulmonary nodules in multi centers: Peking University People's Hospital (200 participants), The First Affiliated Hospital of Zhengzhou University (200 participants), and Beijing Haidian Hospital (100 participants).
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity of breath test combined with computed tomography | 8 weeks
  Using pathological diagnosis of pulmonary nodule as gold standard, diagnostic specificity of breath test combined with computed tomography will be calculated
Diagnostic specificity of breath test combined with computed tomography | 8 weeks
  Using pathological diagnosis of pulmonary nodule as gold standard, diagnostic specificity of breath test combined with computed tomography will be calculated
Diagnostic accuracy of breath test combined with computed tomography | 8 weeks
  Using pathological diagnosis of pulmonary nodule as gold standard, diagnostic accuracy of breath test combined with computed tomography will be calculated

SECONDARY OUTCOMES:
Positive predictive value of breath test combined with computed tomography | 8 weeks
  Using pathological diagnosis of pulmonary nodule as gold standard, positive predictive value of breath test combined with computed tomography will be calculated
Negative predictive value of breath test combined with computed tomography | 8 weeks
  Using pathological diagnosis of pulmonary nodule as gold standard, negative predictive value of breath test combined with computed tomography will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Mantang Qiu, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No